CLINICAL TRIAL: NCT01240746
Title: Safety and Immunogenicity Among Children Administered Quadrivalent Influenza Vaccine
Brief Title: Study of Quadrivalent Influenza Vaccine Among Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QIV04; UTN: U1111-1114-3713 (Other: WHO)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Influenza Vaccine; Trivalent Influenza Vaccine; Influenza viruses; Fluzone®
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Licensed 2010-2011 TIV (Active Comparator): Participants will receive the Licensed 2010-2011 Trivalent Influenza Vaccine containing the primary B strain.
  Interventions: Biological: Licensed 2010-2011 Trivalent Influenza Vaccine, No Preservative
- Group 2: Investigational TIV (Experimental): Participants will receive the Investigational Trivalent Influenza Vaccine containing the alternate B strain
  Interventions: Biological: Investigational Trivalent Influenza Vaccine with alternate B strain, No Preservative
- Group 3: Investigational QIV (Experimental): Participants will receive the investigational Quadrivalent Influenza Vaccine
  Interventions: Biological: Quadrivalent Influenza Vaccine, No Preservative

INTERVENTIONS:
Biological: Licensed 2010-2011 Trivalent Influenza Vaccine, No Preservative — 0.25 mL (6 to 35 months) or 0.5 mL (3 to <9 years), Intramuscular
  Other Names: Fluzone®
  Arms: Group 1: Licensed 2010-2011 TIV
Biological: Investigational Trivalent Influenza Vaccine with alternate B strain, No Preservative — 0.25 mL (6 to 35 months) or 0.5 mL (3 to <9 years), Intramuscular
  Arms: Group 2: Investigational TIV
Biological: Quadrivalent Influenza Vaccine, No Preservative — 0.25 mL (6 to 35 months), or 0.5 mL(3 to <9 years), Intramuscular
  Arms: Group 3: Investigational QIV

SUMMARY:
The aim of the study is to evaluate a prototype quadrivalent influenza vaccine (QIV), the licensed 2010-2011 trivalent influenza vaccine (TIV) containing the primary B strain (B1), and the investigational TIV containing the alternate B (B2) strain in children.

Primary Objective:

To demonstrate non-inferiority of antibody responses to QIV compared with licensed 2010-2011 TIV (containing the primary B strain) and investigational TIV (containing the alternate B strain) as assessed by geometric mean titer (GMT) ratios for each of the four virus strains separately among children aged 6 months to less than 9 years of age

Secondary Objective:

To demonstrate superiority of antibody responses to each B strain in QIV compared with antibody titers following vaccination with the TIV that does not contain the corresponding B strain, as assessed by GMT ratios and seroconversion rates.

Observational Objective:

To describe the safety profile of QIV among subjects 6 months to less than 9 years of age, as assessed by solicited injection site and systemic adverse events (AEs) collected for 7 days post-vaccination, unsolicited adverse events collected from 21 days post-vaccination, and adverse events of special interest and serious adverse events (SAEs) collected from Visit 1 to Visit 2.

DETAILED DESCRIPTION:
Participants will receive a single dose of their assigned vaccine during Visit 1. For those requiring two doses of influenza vaccine, as per Advisory Committee on Immunization Practices (ACIP) guidance, a second dose of the assigned vaccine will be administered at Visit 2. All participants will be followed up for safety (up to 6 months post final vaccination) and for immunogenicity up to Day 28 post-vaccination (Visit 2 or Visit 3, as appropriate).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 6 months to < 9 years of age on the day of inclusion.
* Parent/guardian is willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Subject is in reasonably good health as assessed by the Investigator.
* Informed consent is granted by the parent(s) or other legally acceptable representative; assent by subjects 7 to < 9 years of age.
* For subjects 6 months to < 24 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* History of allergy to egg proteins or any constituents of the vaccine.
* History of serious adverse reaction to any influenza vaccine.
* Any vaccination scheduled between Visit 1 and Visit 2 (or Visit 1 and Visit 3 for those requiring two doses).
* Receipt of any vaccine in the 4 weeks preceding the first study vaccination.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first study vaccination or during the course of the study.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré syndrome.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Personal or immediate family history of congenital immune deficiency.
* Personal developmental delay, neurologic disorder, or seizure disorder.
* Any chronic illness that, in the opinion of the Investigator, is not well controlled and may interfere with trial conduct or completion, or with assessment of adverse events.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.
* Receipt of blood or blood-derived products (including immunoglobulin therapy) in the past 3 months, which might interfere with assessment of the immune response.
* Employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4363 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (58):
- United States (58):
  - Dothan, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - San Diego, California
  - Colorado Spring, Colorado
  - Denver, Colorado
  - Ridgefield, Connecticut
  - Boca Raton, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami Beach, Florida
  - Ponte Vedra, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Marietta, Georgia
  - Arkansas City, Kansas
  - Newton, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Metairie, Louisiana
  - Columbia, Maryland
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Binghamton, New York
  - Cary, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Scranton, Pennsylvania
  - Warwick, Rhode Island
  - Barnwell, South Carolina
  - Mt. Pleasant, South Carolina
  - Clarksville, Tennessee
  - Kingsport, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Katy, Texas
  - Layton, Utah
  - Murray, Utah
  - Orem, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Williamsburg, Virginia
  - Marshfield, Wisconsin

REFERENCES:
- [Result] Greenberg DP, Robertson CA, Landolfi VA, Bhaumik A, Senders SD, Decker MD. Safety and immunogenicity of an inactivated quadrivalent influenza vaccine in children 6 months through 8 years of age. Pediatr Infect Dis J. 2014 Jun;33(6):630-6. doi: 10.1097/INF.0000000000000254. PMID 24445833
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 11 November 2010 to 20 June 2011 in 69 clinical centers in the US
Pre-assignment Details: A total of 4363 participants who met all the inclusion criteria and none of the exclusion criteria were enrolled, randomized and vaccinated in the study.
Groups:
- Study Group 1 (2010-2011 Trivalent Influenza Vaccine): Participants received the Licensed 2010-2011 Trivalent Influenza Vaccine (TIV) containing the primary B strain influenza antigen.
- Study Group 2 (Investigational Trivalent Influenza Vaccine): Participants received the Investigational Trivalent Influenza Vaccine (TIV) containing the alternate B strain influenza antigen
- Study Group 3 (Investigational Quadrivalent Influenza Vaccine): Participants received the Investigational Quadrivalent Influenza Vaccine (QIV)
Period: Overall Study
Arm/Group | Study Group 1 (2010-2011 Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Started | 736 | 725 | 2902
Completed | 677 | 677 | 2659
Not Completed | 59 | 48 | 243
Not completed — Adverse Event | 2 | 0 | 10
Not completed — Lost to Follow-up | 23 | 20 | 102
Not completed — Protocol Violation | 24 | 15 | 72
Not completed — Withdrawal by Subject | 10 | 13 | 59

BASELINE CHARACTERISTICS:
Groups:
- Study Group 1 (Trivalent Influenza Vaccine): Participants received the Licensed 2010-2011 Trivalent Influenza Vaccine (TIV) containing the primary B strain influenza antigen
- Total: Total of all reporting groups
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine) | Total
Number analyzed (Participants) | 736 | 725 | 2902 | 4363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 736 | 725 | 2902 | 4363
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 49.6 (29.0) | 49.6 (28.7) | 49.8 (29.7) | 49.8 (29.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 359 | 1427 | 2153
  Male | 369 | 366 | 1475 | 2210
Region of Enrollment [Number; unit: Participants]
  United States | 736 | 725 | 2902 | 4363

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers Against Influenza A Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Participants
Description: Immunogenicity outcomes were assessed in serum samples by hemagglutination inhibition (HAI) assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: Day 28 post final vaccination
Population: Geometric mean titers (GMT) to influenza vaccine A antigens were determined in randomized and vaccinated participants, per-protocol population. The GMT data for antigen A/Victoria/210/2009 and A/California/07/2009 were pooled for participants vaccinated with either 2010-2011 TIV or the investigational TIV. Data presented in column for Group 1.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 1461 | 0 | 2339
Titers
  A/California/07/2009 (A/H1N1) [N = 1461, 0, 2339] | 1096 [1008 to 1192] |  | 1124 [1060 to 1192]
  A/Victoria/210/2009 (A/H3N2) [N = 1461, 0, 2339 | 828 [774 to 887] |  | 822 [783 to 862]

2. Other Pre Specified Outcome: Seroconversion Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines With Corresponding B Strain in All Participants
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroconversion was defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and ≥four-fold increase in post-vaccination
Time Frame: Day 28 post final vaccination
Population: Seroconversion with respect to influenza vaccine B antigens were determined in randomized and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Participants
  B/Brisbane/60/2008 (581, 0, 2336) | 355 | NA [0 to 0] — B/Brisbane/60/2008 antigen was not in the influenza vaccine administered to this group. | 1677 [0 to 0]
  B/Florida/04/2006 (0, 598, 2335) | NA — B/Florida/04/2006 antigen was not in the influenza vaccine administered to this group. | 383 [0 to 0] | 1543 [0 to 0]

3. Primary Outcome: Geometric Mean Titers Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines With Corresponding B Strain in All Participants
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
Time Frame: Day 28 post final vaccination
Population: Geometric mean titers to influenza vaccine B antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the B antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Titers
  B/Brisbane/60/2008 (581, 0, 2238) | 64.3 [58.3 to 70.9] | NA [NA to NA] — B/Brisbane/60/2008 antigen was not in the influenza vaccine administered to this group. | 86.1 [81.8 to 90.6]
  B/Florida/04/2006 (0, 598, 2338) | NA [NA to NA] — B/Florida/04/2006 antigen was not in the influenza vaccine administered to this group. | 58.3 [52.6 to 64.7] | 61.5 [58.6 to 64.7]

4. Primary Outcome: Geometric Mean Titers Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines Without Corresponding B Strain in All Participants
Description: as for outcome 3
Time Frame: Day 28 post final vaccination
Population: Geometric mean titers to influenza vaccine B antigens (cross-reactive antibody) were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the B antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Titers
  B/Brisbane/60/2008 (0, 599, 2338) | NA [NA to NA] — B/Florida/04/2006 antigen was not in the influenza vaccine administered to this group. | 19.5 [17.4 to 21.8] | 86.1 [81.8 to 90.6]
  B/Florida/04/2006 (581, 0, 2338) | 16.3 [14.8 to 17.9] | NA [NA to NA] — B/Brisbane/60/2008 antigen was not in the influenza vaccine administered to this group. | 61.5 [58.6 to 64.7]

5. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Participants
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroprotection was defined as a pre-vaccination and post-vaccination titer ≥ 40 (l/dil)
Time Frame: Day 28 post final vaccination
Population: Seroprotection against influenza vaccine antigens was determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the particular antigen.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Participants
  A/H1N1 Pre-vaccination (581, 599, 2333) | 291 | 305 [0 to 0] | 1159 [0 to 0]
  A/H1N1 Post-vaccination (581, 597, 2337) | 573 | 585 [0 to 0] | 2305 [0 to 0]
  A/H3N2 Pre-vaccination (579, 596, 2334) | 248 | 241 [0 to 0] | 946 [0 to 0]
  A/H3N2 Post-vaccination (580, 599, 2334) | 575 | 593 [0 to 0] | 2326 [0 to 0]
  B/Brisbane Pre-vaccination 582, 599, 2337) | 64 | 79 [25.0 to 33.7] | 261 [0 to 0]
  B/Brisbane Post-vaccination (581, 599, 2338) | 418 | 202 [0 to 0] | 1838 [0 to 0]
  B/Florida Pre-vaccination (582, 598, 2336) | 51 | 55 [0 to 0] | 199 [0 to 0]
  B/Florida Post-vaccination (581, 598, 2338) | 169 | 416 [0 to 0] | 1674 [0 to 0]

6. Other Pre Specified Outcome: Seroconversion Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Participants
Description: Immunogenicity outcomes were assessed in serum samples by HAI assay. The lower limit of quantitation (LLOQ) was set at the lowest dilution used in the assay, 1/10. Titers below this level were reported as <10.
  Seroconversion was defined as either a pre vaccination HAI titer <1:10 and a post vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and a four-fold increase in post-vaccination.
Time Frame: Day 28 post final vaccination
Population: Seroconversion with respect to vaccine antigens (cross-reactive antibody) were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the particular antigen.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Participants
  A/H1N1 (580, 597, 2331) | 541 | 535 [0 to 0] | 2135 [0 to 0]
  A/H3N2 (578, 596, 2329) | 477 | 512 [0 to 0] | 2050 [0 to 0]
  B/Brisbane (581, 599, 2336) | 355 | 120 [0 to 0] | 1677 [0 to 0]
  B/Florida (581, 598, 2335) | 104 | 383 [0 to 0] | 1543 [0 to 0]

7. Primary Outcome: Geometric Mean Titers Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in Participants Aged 6 Months to Less Than 36 Months.
Description: as for outcome 3
Time Frame: Day 28 post final vaccination
Population: Geometric mean titers to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants aged 6 months to less than 36 months with valid serology results for the particular antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 225 | 245 | 949
Titers
  A/H1N1, Pre-vaccination (224, 245, 943) | 25.6 [19.4 to 33.7] | 31.3 [23.8 to 41.1] | 25.7 [22.4 to 29.5]
  A/H1N1, Post-vaccination (224, 243, 947) | 797 [664 to 957] | 645 [530 to 784] | 747 [680 to 821]
  A/H3N2, Pre-vaccination (224, 245, 945) | 9.52 [7.90 to 11.5] | 10.1 [8.26 to 12.3] | 9.19 [8.42 to 10.0]
  A/H3N2, Post-vaccination (224, 243, 944) | 558 [483 to 646] | 583 [507 to 671] | 526 [492 to 562]
  B/Brisbane, Pre-vaccination (225, 245, 947) | 6.56 [5.92 to 7.27] | 6.62 [6.00 to 7.30] | 6.41 [6.10 to 6.73]
  B/Brisbane, Post-vaccination (225, 245, 948) | 54.7 [47.2 to 63.4] | 12.0 [10.3 to 13.9] | 72.8 [67.3 to 78.7]
  B/Florida, Pre-vaccination (225, 245, 946) | 5.33 [5.10 to 5.56] | 5.26 [5.09 to 5.44] | 5.34 [5.23 to 5.46]
  B/Florida, Post-vaccination (225, 245, 948) | 8.56 [7.68 to 9.54] | 32.9 [28.7 to 37.6] | 36.2 [33.7 to 38.8]

8. Other Pre Specified Outcome: Seroconversion Against Influenza B Strains After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines Without Corresponding B Strain in All Participants.
Description: as for outcome 6
Time Frame: Day 28 post final vaccination
Population: Seroconversion with respect to influenza vaccine B antigens (cross-reactive antibody) was determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the B antigens.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 582 | 599 | 2339
Participants
  B/Brisbane/60/2008 (0, 599, 2336) | NA — B/Florida/04/2006 antigen was not in the influenza vaccine administered to this group | 120 | 1677
  B/Florida/04/2006 (581, 0, 2335) | 104 | NA — B/Brisbane/60/2008 antigen was not in the influenza vaccine administered to this group | 1543

9. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in Participants Aged 6 Months to Less Than 36 Months.
Description: as for outcome 5
Time Frame: Day 28 post final vaccination
Population: Seroprotection against influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants aged 6 months to less than 36 months with valid serology results for the particular antigen.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 225 | 245 | 949
Participants
  H1N1 Pre-vaccination (224, 245, 943) | 80 | 100 | 327
  H1N1 Post-vaccination (223, 243, 941) | 220 | 237 | 925
  H3N2 Pre-vaccination (224, 245, 945) | 26 | 29 | 104
  H3N2 Post-vaccination (223, 243, 944) | 221 | 242 | 943
  B/Brisbane Pre-vaccination (225, 245, 947) | 14 | 18 | 61
  B/Brisbane Post-vaccination (225, 245, 948) | 155 | 55 | 716
  B/Florida Pre-vaccination (225, 245, 946) | 4 | 1 | 10
  B/Florida Post-vaccination (225, 245, 948) | 19 | 135 | 550

10. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in Participants Aged 3 Years to Less Than 9 Years.
Description: as for outcome 5
Time Frame: Day 28 post-vaccination
Population: Seroprotection against influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants aged 3 years to less than 9 years with valid serology results for the particular antigen.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 357 | 354 | 1390
Participants
  H1N1 Pre-vaccination (357, 354, 1390) | 211 | 205 | 832
  H1N1 Post-vaccination (357, 354, 1390) | 353 | 348 | 1380
  H3N2 Pre-vaccination (355, 353, 1389) | 222 | 212 | 842
  H3N2 Post-vaccination (356, 353, 1390) | 354 | 351 | 1383
  B/Brisbane Pre-vaccination (357, 354, 1390) | 50 | 61 | 200
  B/Brisbane Post-vaccination (356, 354, 1390) | 263 | 147 | 1122
  B/Florida Pre-vaccination (357, 353, 1390) | 47 | 54 | 189
  B/Florida Post-vaccination (356, 353, 1390) | 150 | 281 | 1124

11. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With One Dose of Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Participants
Description: as for outcome 5
Time Frame: Day 28 post-vaccination
Population: Seroprotection against influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants with valid serology results for the particular antigen.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 114 | 141 | 510
Participants
  H1N1 Pre-vaccination (114, 141, 510) | 62 | 89 | 289
  H1N1 Post-vaccination (114, 141, 510) | 111 | 139 | 498
  H3N2 Pre-vaccination (112, 141, 510) | 64 | 75 | 259
  H3N2 Post-vaccination (112, 141, 510) | 110 | 138 | 504
  B/Brisbane Pre-vaccination (114, 141, 510) | 15 | 25 | 66
  B/Brisbane Post-vaccination (113, 141, 510) | 72 | 55 | 341
  B/Florida Pre-vaccination (114, 141, 510) | 18 | 20 | 58
  B/Florida Post-vaccination (113, 141, 510) | 46 | 98 | 350

12. Other Pre Specified Outcome: Seroprotection Against Influenza Vaccine Antigens After Vaccination With Two Doses of Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in All Participants
Description: as for outcome 5
Time Frame: Day 28 post final vaccination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 468 | 458 | 1829
Participants
  H1N1 Pre-vaccination (467, 458, 1823) | 229 | 216 | 870
  H1N1 Post-vaccination (467, 456, 1827) | 462 | 446 | 1807
  H3N2 Pre-vaccination (467, 457, 1824) | 184 | 166 | 687
  H3N2 Post-vaccination (467, 455, 1824) | 465 | 455 | 1822
  B/Brisbane Pre-vaccination (468, 458, 1827) | 49 | 54 | 195
  B/Brisbane Post-vaccination (468, 458, 1828) | 346 | 147 | 1497
  B/Florida Pre-vaccination (468, 457, 1826) | 33 | 35 | 141
  B/Florida Post-vaccination (468, 457, 1828) | 123 | 318 | 1324

13. Primary Outcome: Geometric Mean Titers Against Influenza Vaccine Antigens After Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines in Participants Aged 3 Years to Less Than 9 Years.
Description: as for outcome 3
Time Frame: Day 28 post-vaccination
Population: Geometric mean titers to influenza vaccine antigens were determined in randomized and vaccinated participants, per-protocol population. Data presented for participants aged 3 years to less than 9 Years with valid serology results for the particular antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 357 | 354 | 1390
Titers
  A/H1N1, Pre-vaccination (357, 354, 1390) | 53.5 [43.9 to 65.2] | 54.4 [44.4 to 66.8] | 54.9 [49.6 to 60.7]
  A/H1N1, Post-vaccination (357, 354, 1390) | 1565 [1355 to 1807] | 1348 [1166 to 1559] | 1484 [1380 to 1595]
  A/H3N2, Pre-vaccination (355, 353, 1389) | 70.6 [57.3 to 87.0] | 64.1 [51.9 to 79.2] | 63.9 [57.6 to 70.8]
  A/H3N2, Post-vaccination (356, 353, 1390) | 924 [816 to 1046] | 1214 [1078 to 1367] | 1112 [1046 to 1183]
  B/Brisbane, Pre-vaccination (357, 354, 1390) | 10.1 [9.05 to 11.2] | 10.6 [9.52 to 11.9] | 9.73 [9.23 to 10.3]
  B/Brisbane, Post-vaccination (356, 354, 1390) | 71.2 [62.6 to 81.1] | 27.3 [23.4 to 31.8] | 96.6 [90.3 to 103]
  B/Florida, Pre-vaccination (357, 353, 1390) | 9.09 [8.26 to 10.0] | 9.84 [8.91 to 10.9] | 9.34 [8.89 to 9.82]
  B/Florida, Post-vaccination (356, 353, 1390) | 24.4 [21.6 to 27.5] | 86.9 [76.1 to 99.2] | 88.5 [83.1 to 94.1]

14. Other Pre Specified Outcome: Number of Participants Aged 6 Months to <36 Months Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines.
Description: Solicited injection site reactions (Age 6-23 Months): Tenderness, Erythema and Swelling. Solicited systemic reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability.
  Grade 3: Tenderness: cries when injected limb is moved; Erythema and Swelling ≥ 50 mm; Fever: >103.1°F; Vomiting: ≥6 episodes/24 hours; Abnormal crying: >3 hours; Drowsiness: Sleeping most of the time; Loss of appetite: refuses ≥3 feeds/meals or most feeds/meals; Irritability: inconsolable.
  Solicited Injection site reactions (Age 24 Months to < 36 months): Pain, Erythema, and Swelling. Systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
  Grade 3: Pain: Incapacitating, unable to perform usual activities; Redness and Swelling: ≥ 50 mm; Fever: ≥102.1°F; Headache, Malaise and Myalgia: Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety profile were assessed in all randomized and vaccinated participants, safety population. Values presented for participants aged 6 months to <36 months with available data for the relevant endpoint.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 310 | 308 | 1223
Participants
  Injection site Pain (130, 149, 521) | 68 | 75 [0 to 0] | 297 [0 to 0]
  Grade 3 Injection site Pain (130, 149, 521) | 1 | 4 [0 to 0] | 5 [0 to 0]
  Injection site Tenderness (159, 145, 628) | 77 | 72 | 340
  Grade 3 Injection site Tenderness (159, 145, 628) | 3 | 0 | 12
  Injection site Erythema (289, 294, 1150) | 95 | 98 [0 to 0] | 429 [0 to 0]
  Grade 3 Injection site Erythema (289, 294, 1150) | 0 | 0 [0 to 0] | 2 [0 to 0]
  Injection site Swelling (289, 294, 1150) | 57 | 51 [0 to 0] | 248 [0 to 0]
  Grade 3 Injection site Swelling (289, 294, 1150) | 0 | 0 [0 to 0] | 2 [0 to 0]
  Fever (288, 293, 1148) | 46 | 38 [0 to 0] | 164 [0 to 0]
  Grade 3 Fever (288, 293, 1148) | 5 | 6 [0 to 0] | 24 [0 to 0]
  Vomiting (159, 144, 628) | 18 | 20 | 93
  Grade 3 Vomiting (159, 144, 628) | 1 | 0 | 6
  Crying abnormal (159, 144, 628) | 58 | 43 | 259
  Grade 3 Crying abnormal (159, 144, 628) | 3 | 3 | 21
  Drowsiness (159, 144, 628) | 51 | 46 | 237
  Grade 3 Drowsiness (159, 144, 628) | 1 | 1 | 8
  Headache (128, 148, 517) | 12 | 18 [0 to 0] | 46 [0 to 0]
  Grade 3 Headache (128, 148, 517) | 0 | 0 [0 to 0] | 3 [0 to 0]
  Appetite lost (159, 144, 628) | 53 | 36 | 203
  Grade 3 Appetite lost (159, 144, 628) | 3 | 1 | 11
  Malaise (128, 148, 517) | 45 | 48 [0 to 0] | 197 [0 to 0]
  Grade Malaise (128, 148, 517) | 6 | 10 [0 to 0] | 24 [0 to 0]
  Myalgia (128, 148, 517) | 34 | 37 [0 to 0] | 138 [0 to 0]
  Grade 3 Myalgia (128, 148, 517) | 2 | 4 [0 to 0] | 10 [0 to 0]
  Irritability (159, 144, 628) | 84 | 77 | 339
  Grade 3 Irritability (159, 144, 628) | 5 | 4 | 20

15. Other Pre Specified Outcome: Number of Participants Aged 3 Years to <9 Years Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Fluzone® Quadrivalent Influenza Vaccine or Trivalent Influenza Vaccines
Description: Solicited injection site reactions: Pain, Redness, and Swelling. Solicited systemic reactions: Fever (Temperature); Headache, Malaise and Myalgia Grade 3 Pain: incapacitating, unable to perform usual activities; Redness and Swelling: ≥ 50 mm; Fever: ≥ 102.1°F; Headache, Malaise and Myalgia: Significant, prevents daily activity, respectively.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety profile were assessed in all randomized and vaccinated participants, safety population. Values presented for participants aged 3 years to <9 years with available data for the relevant endpoint.
Measure: Number; unit: Participants
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Number analyzed (Participants) | 424 | 413 | 1669
Participants
  Injection site Pain (410, 398, 1592) | 265 | 254 | 1061
  Grade 3 Injection site Pain (410, 398, 1592) | 8 | 11 | 33
  Injection site Erythema (410, 398, 1592) | 151 | 140 | 543
  Grade 3 Injection site Erythema (410, 398, 1592) | 5 | 7 | 29
  Injection site Swelling (410, 398, 1592) | 104 | 103 | 395
  Grade 3 Injection site Swelling (410, 398, 1592) | 5 | 7 | 22
  Fever (409, 396, 1591) | 29 | 30 | 112
  Grade 3 Fever (409, 396, 1591) | 5 | 3 | 34
  Headache (411, 398, 1593) | 87 | 97 | 368
  Grade 3 Headache (411, 398, 1593) | 11 | 8 | 35
  Malaise (411, 398, 1593) | 135 | 133 | 508
  Grade 3 Malaise (411, 398, 1593) | 23 | 20 | 87
  Myalgia (411, 398, 1593) | 140 | 153 | 615
  Grade 3 Myalgia (411, 398, 1593) | 11 | 11 | 52

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 (post-vaccination) up to 6 months post-vaccination.
Description: Data are presented for participants with available safety data for the relevant endpoints.
Arm/Group | Study Group 1 (Trivalent Influenza Vaccine) | Study Group 2 (Investigational Trivalent Influenza Vaccine) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine)
Serious Adverse Events (participants affected / at risk) | 7/734 | 14/721 | 41/2892
Other Adverse Events (participants affected / at risk) | 333/734 | 329/721 | 1358/2892
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Group 1 (Trivalent Influenza Vaccine) (N=734) | Study Group 2 (Investigational Trivalent Influenza Vaccine) (N=721) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine) (N=2892)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Drowning (General disorders) | 1/225 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Respiratory syncytial vrus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Respiratory syncytial vrus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (10)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Autism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2) | 3 (3) | 8 (8)
Seizure anoxic (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (8)
Bronchial hrperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Study Group 1 (Trivalent Influenza Vaccine) (N=734) | Study Group 2 (Investigational Trivalent Influenza Vaccine) (N=721) | Study Group 3 (Investigational Quadrivalent Influenza Vaccine) (N=2892)
Injection site pain (General disorders) | 333/540 (333) | 329/547 (329) | 1358/2113 (1358)
Injection site Swelling (General disorders) | 161 (162) | 154/692 (154) | 643/2742 (643)
Headache (Nervous system disorders) | 99/539 (99) | 115/546 (115) | 414/2110 (414)
Malaise (General disorders) | 180/539 (180) | 181/546 (181) | 705/2110 (705)
Myalgia (Musculoskeletal and connective tissue disorders) | 174/539 (174) | 190/546 (190) | 753/2110 (753)
Injection site tenderness (General disorders) | 77/159 (77) | 72/145 (72) | 340/628 (340)
Injection site erythema (General disorders) | 246/699 (246) | 238/692 (238) | 972/2742 (972)
Fever (General disorders) | 75/695 (75) | 68/689 (68) | 276/2739 (276)
Vomiting (Gastrointestinal disorders) | 18/159 (18) | 20/144 (20) | 93/628 (93)
Appetite lost (Metabolism and nutrition disorders) | 53/159 (53) | 36/144 (36) | 203/628 (203)
Drowsiness (Nervous system disorders) | 51/159 (51) | 46/144 (46) | 237/628 (237)
Crying abnormal (Psychiatric disorders) | 58/159 (58) | 43/144 (43) | 259/628 (259)
Irritability (Psychiatric disorders) | 84/159 (84) | 77/144 (77) | 339/628 (339)
Diarrhoea (Gastrointestinal disorders) | 42 (51) | 38 (48) | 135 (150)
Vomiting (Gastrointestinal disorders) | 46 (52) | 55 (61) | 193 (209)
Pyrexia (General disorders) | 44 (49) | 65 (75) | 188 (213)
Upper respiratory tract infection (Infections and infestations) | 43 (51) | 47 (50) | 184 (203)
Cough (Respiratory, thoracic and mediastinal disorders) | 95 (107) | 89 (100) | 341 (381)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 37 (38) | 34 (39) | 167 (189)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.